CLINICAL TRIAL: NCT04168554
Title: Pilotonderzoek Naar Het Gebruik Van Telemedicine Bij Het Beoordelen Van Het Benauwde Kind in de Huisartsenpraktijk English: The Use of Telemedicine in the General Practitioners Office for a Child With Respiratory Symptoms: a Pilot Study
Brief Title: Telemedicine in the Generals Practitioners Office
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1384
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Distress Syndrome; Pneumonia; Bronchiolitis; Croup; Croup; False; Asthma; Bronchial Hyperreactivity
Keywords: Telemedicine; Respiratory distress; Pediatric; General practitioner
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Bronchiolitis; Croup; Asthma; Bronchial Hyperreactivity; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Phase 1 and Phase 2: 20 patients studied in the emergency room with a pediatrician not presen in the ER performing the telemedicine examination from a distance (ie an office down the hall) followed directly by a face-to-face
  20 patients included in the general practitioners office, telemedicine is performed from within the hospital to the GPs office.
  Patient is then still referred to the hospital in order to check whether the telemedicine and face-to-face examination are somewhat similarce physical examination
  Interventions: Device: Telemedicine

INTERVENTIONS:
Device: Telemedicine — Patient is examined using telemedicine

SUMMARY:
Pediatrician does physical examination through telemedicine and in real life to see whether the telemedicine consultation corresponds with the real life examination.

Goal is to determine:

1. Check practical feasability
2. Check whether there are no great objections for a larger study (ie. in case telemedicine consultation is much more unreliable to do a physical examination a larger study is deemed unsafe)

DETAILED DESCRIPTION:
40 pediatric patients seen by a general practitioner (GP) whom the GP has referred or wants to refer to a pediatrician for clinical evaluation are included in this study.

Study is designed in 2 parts. Part 1 is at the emergency room in the hospital Part 2 is at the GPs office

The pediatrician sees the patient through a telemedicine consultation. Then sees the patient in real life to see if what was seen during telemedicine corresponds with the real life consultation.

With telemedicine and real life consultation the pediatrician rates the patient as either a candidate to go home or to be admitted. With the telemedicine consultation there is also an option "in doubt: i want to see the patient in real life".

Also with both telemedicine and real life examination the pediatrician scores the patient using the respiratory observation scale (Siew et al, 2016)

Goal is to:

1. Check practical feasability
2. Check whether there are no great objections for a larger study (ie. in case telemedicine consultation is much harder to do a physical examination

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with respiratory symptoms whom are referred by a general practitioner to be evaluated by a pediatrician

Exclusion Criteria:

* Infants younger than 2 months of age
* 19 years and older
* Ex-premature with post-conceptional age <48 weeks
* Congenital heart disease
* Down Syndrome
* Immune deficiency
* Pre-existent pulmonary disorder (Broncho-pulmonary dysplasia, Cystic Fibrosis)
* Pre-existent neurological disorders
* Apnea's
* Patients with respiratory distress with dehydration symptoms
* Patients who have already been treated with salbutamol inhalers of nebulizer - Emergency patient with respiratory insufficiency
* Technical problems which cause a delay longer than 10 minutes before a video-connection is made
* expected delay before commencing telemedicine consultation of longer than 30 minutes

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with any type of respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Discharge or admitted? | within 30-60 minutes after inclusion
  Patients are categorized in one of three categories through telemedicine-evaluation Group 1: "Patient can safely go home" Group 2: "Patient will need to be admitted" Group 3: "In doubt between group 1 and group 2, emergency room consultation required" FTF evaluation: Group 1: "Patient can safely go home" Group 2: "Patient will need to be admitted"
Respiratory Observation Scale | within 30-60 minutes after inclusion
  Observe the presence of: tachypnea, nasal flaring, perioral cyanosis, tripoding, thoracoabdominal asynchrony, supraclavicular-, substernal- or intercostal retractions, mental status and patient in respiratory distress

SECONDARY OUTCOMES:
Patient reported experience measure | within 60 minutes after telemedicine evaluation
  questionnaire on patient / parent satisfaction with regard to the telemedicine
Doctor reported experience measure | within 4 weeks after inclusion of patients
  Interview with participating doctors with regard to satisfaction of the telemedicine

CONTACTS AND LOCATIONS:
Overall Officials: Margreet Wessels, MD, PhD, Principal Investigator — Rijnstate Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siew L, Hsiao A, McCarthy P, Agarwal A, Lee E, Chen L. Reliability of Telemedicine in the Assessment of Seriously Ill Children. Pediatrics. 2016 Mar;137(3):e20150712. doi: 10.1542/peds.2015-0712. Epub 2016 Feb 5. PMID 26908666